CLINICAL TRIAL: NCT04134728
Title: A 24-week, Phase 3, Multicentre, Randomised, Double-blind, Efficacy and Safety Study, Comparing GSK3196165 With Placebo and With Sarilumab, in Combination With Conventional Synthetic DMARDs, in Participants With Moderately to Severely Active Rheumatoid Arthritis Who Have an Inadequate Response to Biological DMARDs and/or Janus Kinase Inhibitors
Brief Title: Efficacy and Safety of GSK3196165 (Otilimab) Versus Placebo and Sarilumab in Participants With Moderately to Severely Active Rheumatoid Arthritis Who Have an Inadequate Response to Biological Disease-modifying Antirheumatic Drug (DMARDs) and/or Janus Kinase (JAK) Inhibitors
Acronym: contRAst 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202018
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Arthritis, Rheumatoid
Keywords: bDMARD; GSK3196165; Rheumatoid Arthritis; Sarilumab; Otilimab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Otilimab; sarilumab

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of six intervention arms in ratio of 6:6:6:1:1:1
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- GSK3196165 90 mg (Experimental): Entire treatment period (24 Weeks): GSK3196165 90 mg SC injection once weekly. Participants will also receive a stable dose of csDMARD(s) as standard of care (SoC).
  Interventions: Biological: GSK3196165 (Otilimab); Drug: csDMARDs
- GSK3196165 150 mg (Experimental): Entire treatment period (24 Weeks): GSK3196165 150 mg SC injection once weekly. Participants will also receive a stable dose of csDMARD(s) as SoC.
  Interventions: Biological: GSK3196165 (Otilimab); Drug: csDMARDs
- Sarilumab 200 mg (Active Comparator): Entire treatment period (24 Weeks): Sarilumab 200 mg SC injection every other week + placebo SC injection in the intervening weeks. Participants will also receive a stable dose of csDMARD(s) as SoC.
  Interventions: Biological: Sarilumab; Drug: Placebo to GSK3196165/ Sarilumab; Drug: csDMARDs
- Placebo sequence 1 (Placebo Comparator): From Week 0-11: Placebo SC injection once weekly. From Week 12 onwards: GSK3196165 90 mg SC injection once weekly. Participants will also receive a stable dose of csDMARD(s) as SoC.
  Interventions: Biological: GSK3196165 (Otilimab); Drug: Placebo to GSK3196165/ Sarilumab; Drug: csDMARDs
- Placebo sequence 2 (Placebo Comparator): From Week 0-11: Placebo SC injection once weekly. From Week 12 onwards: GSK3196165 150 mg SC injection once weekly. Participants will also receive a stable dose of csDMARD(s) as SoC.
  Interventions: Biological: GSK3196165 (Otilimab); Drug: Placebo to GSK3196165/ Sarilumab; Drug: csDMARDs
- Placebo sequence 3 (Placebo Comparator): From Week 0-11: Placebo SC injection once weekly. From Week 12 onwards: Sarilumab 200 mg SC injection every other week + placebo SC injection in the intervening weeks. Participants will also receive a stable dose of csDMARD(s) as SoC.
  Interventions: Biological: Sarilumab; Drug: Placebo to GSK3196165/ Sarilumab; Drug: csDMARDs

INTERVENTIONS:
Biological: GSK3196165 (Otilimab) — GSK3196165 solution in vial/pre-filled syringe (PFS) to be administered SC.
  Arms: GSK3196165 150 mg; GSK3196165 90 mg; Placebo sequence 1; Placebo sequence 2
Biological: Sarilumab — Sarilumab solution in PFS to be administered SC.
  Arms: Placebo sequence 3; Sarilumab 200 mg
Drug: Placebo to GSK3196165/ Sarilumab — Placebo sterile 0.9 percentage (%) weight by volume (w/v) sodium chloride solution in vial/PFS to be administered SC.
  Arms: Placebo sequence 1; Placebo sequence 2; Placebo sequence 3; Sarilumab 200 mg
Drug: csDMARDs — Stable dose of csDMARD(s) as SoC.

SUMMARY:
This study (contRAst 3 [202018: NCT04134728]) is a Phase 3, randomized, multicenter, double-blind study to assess the safety and efficacy of GSK3196165 in combination with conventional (cs) DMARD[s]) or the treatment of adult participants with moderate to severe active rheumatoid arthritis (RA) who have had an inadequate response to biologic (b) DMARD[s]) and/or JAK inhibitors. The study will consist of a screening phase of up to 6 weeks followed by 24 week treatment phase in which participants will be randomized in ratio of 6:6:6:1:1:1 to GSK3196165 150 milligrams (mg) subcutaneously (SC) weekly,GSK3196165 90 mg SC weekly, sarilumab 200 mg SC every other week or placebo (three arms) respectively, all in combination with background csDMARD(s). At Week 12, participants in the three placebo arms will switch from placebo to active intervention (either GSK3196165 150 mg SC weekly, GSK3196165 90 mg SC weekly, or sarilumab 200 mg SC every other week). Participants who, in investigator's judgement will benefit from extended treatment with GSK3196165, may be included in the long-term extension study (contRAst X [209564: NCT04333147]). Any participant who does not transition into study 209564 will undergo a safety follow-up visit at Week 34 (corresponding to 12 weeks after the last potential dose of sarilumab, at Week 22).

ELIGIBILITY:
Key inclusion criteria:

* >=18 years of age
* Has had RA for >=6 months and was not diagnosed before 16 years of age
* Has active disease, as defined by having both:*

  * >=6/68 tender/painful joints (tender joint count [TJC]), and
  * >=6/66 swollen joints (swollen joint count [SJC])
* Has had an inadequate response despite currently taking at least one and at the most two concomitant csDMARDs for at least 12 weeks, from the following:

  * Methotrexate (MTX)
  * Hydroxychloroquine or chloroquine
  * Sulfasalazine
  * Leflunomide
  * Bucillamine
  * Iguratimod
  * Tacrolimus
* Has had inadequate response to at least one bDMARD at an approved dose and/or at least one JAK inhibitors at an approved dose. In both cases this may be with or without combination with a csDMARD.

  * If surgical treatment of a joint has been performed, that joint cannot be counted in the TJC or SJC.

Key exclusion criteria:

* Has had any active and/or recurrent infections (excluding recurrent fungal infections of the nail bed) or has required management of acute or chronic infections.
* Has received prior treatment with an antagonist of GM-CSF or its receptor.
* Has known infection with human immunodeficiency virus (HIV) or current acute or chronic hepatitis B and/or hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (106):
- United States (39):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Sun City, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Covina, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Tujunga, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Whittier, California
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, DeBary, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Newnan, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Skokie, Illinois
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Minot, North Dakota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Baytown, Texas
  - GSK Investigational Site, College Station, Texas
  - GSK Investigational Site, Colleyville, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lubbock, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, San Marcos, Texas
  - GSK Investigational Site, The Woodlands, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Waco, Texas
- Argentina (8):
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Palta, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, San Isidro, Buenos Aires
  - GSK Investigational Site, San Nicolás de los Arroyos, Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, San Juan
- GSK Investigational Site, Mons, Belgium
- Canada (3):
  - GSK Investigational Site, Barrie, Ontario
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Trois-Rivières, Quebec
- Czechia (5):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Uherské Hradiště
  - GSK Investigational Site, Zlín
- Germany (3):
  - GSK Investigational Site, Rendsburg, Schleswig-Holstein
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Magdeburg
- Hungary (3):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Székesfehérvár
  - GSK Investigational Site, Veszprém
- GSK Investigational Site, Verona, Veneto, Italy
- Japan (14):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
- Lithuania (2):
  - GSK Investigational Site, Klaipėda
  - GSK Investigational Site, Šiauliai
- Poland (12):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Sochaczew
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- South Africa (6):
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Durban, KwaZulu-Natal
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Kempton Park
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Stellenbosch
- South Korea (2):
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
- Spain (5):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Elche
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
- United Kingdom (2):
  - GSK Investigational Site, Romford, Essex
  - GSK Investigational Site, Northwood, Middlesex

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Taylor PC, Weinblatt ME, McInnes IB, Atsumi T, Strand V, Takeuchi T, Bracher M, Brooks D, Davies J, Goode C, Gupta A, Mukherjee S, O'Shea C, Saurigny D, Schifano LA, Shelton C, Smith JE, Wang M, Wang R, Watts S, Fleischmann RM. Anti-GM-CSF otilimab versus sarilumab or placebo in patients with rheumatoid arthritis and inadequate response to targeted therapies: a phase III randomised trial (contRAst 3). Ann Rheum Dis. 2023 Dec;82(12):1527-1537. doi: 10.1136/ard-2023-224449. Epub 2023 Sep 11. PMID 37696589
- See also: 209564 contRAst X NCT04333147 — https://clinicaltrials.gov/ct2/show/NCT04333147?term=209564&draw=2&rank=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized in a ratio of 6:6:6:1:1:1 to GSK3196165 90 milligram (mg):GSK3196165 150mg:Sarilumab:Placebo:Placebo:Placebo. At Week 12, participants randomized to one of the three placebo arms switched to active intervention arms (either GSK3196165 150mg, GSK3196165 90mg or Sarilumab), receiving the active intervention for 12 weeks. Participants randomized to 90mg, GSK3196165 150mg or Sarilumab from study day 1, received the active intervention for 24 weeks.
Pre-assignment Details: Analysis of this study were reported for GSK3196165 90mg, GSK3196165 150mg, Sarilumab and all placebo arms are pooled till Week 12 to primarily serve as reference for comparison of active treatment arms versus Placebo for efficacy objectives at Week 12. Total 550 participants were randomized and one participant from 90mg GSK3196165 withdrew before receiving active intervention due to Protocol Deviation. Hence the participant was removed from intent-to-treat (ITT) and safety population (N=549).
Groups:
- GSK3196165 90mg + csDMARD: Participants between the ages of greater than or equal to (>=)18 years and less than or equal to (<=)84 years received GSK3196165 90 mg + csDMARD administered by weekly subcutaneous injection.
- GSK3196165 150mg + csDMARD: Participants between the ages of greater than or equal to (>=)18 years and less than or equal to (<=)84 years received GSK3196165 150 mg + csDMARD administered by weekly subcutaneous injection.
- Sarilumab 200mg + csDMARD: Participants between the ages of greater than or equal to (>=)18 years and less than or equal to (<=)84 years received Sarilumab 200 mg + csDMARD administered by subcutaneous injection of sarilumab every other week plus with placebo injection in the intervening weeks to maintain the blind.
- Placebo + csDMARD and GSK3196165 90mg + csDMARD: Participants between the ages of greater than or equal to (>=)18 years and less than or equal to(<=)84 years received Placebo +csDMARD until Week 12 later switched toGSK3196165 90 mg +csDMARD administered by weekly subcutaneous injection.
- Placebo + csDMARD and GSK3196165 150mg + csDMARD: Participants between the ages of greater than or equal to (>=)18 years and less than or equal to (<=)84 years received Placebo + csDMARD until Week 12 later switched to GSK3196165 150 mg + csDMARD administered by weekly subcutaneous injection.
- Placebo + csDMARD and Sarilumab 200mg + csDMARD: Participants between the ages of greater than or equal to (>=)18 years and less than or equal to (<=)84 years received Placebo + csDMARD until Week 12 later switched to Sarilumab 200mg + csDMARD administered by subcutaneous injection of sarilumab every other week plus with placebo injection in the intervening weeks to maintain the blind.
Period: Overall Study
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Started | 156 | 158 | 156 | 26 | 26 | 27
Completed | 143 | 144 | 133 | 23 | 25 | 26
Not Completed | 13 | 14 | 23 | 3 | 1 | 1
Not completed — Adverse Event | 3 | 2 | 9 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 3 | 1 | 2 | 0 | 0
Not completed — Protocol-Specified Withdrawal Criterion Met | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Informed Consent Withdrawn | 3 | 6 | 8 | 1 | 1 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1 | 0 | 0 | 1
Not completed — Investigator Site Closed | 0 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD | Total
Number analyzed (Participants) | 156 | 158 | 156 | 26 | 26 | 27 | 549
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 56.7 (10.59) | 56.0 (10.52) | 57.5 (10.69) | 51.6 (11.19) | 57.3 (8.99) | 57.6 (10.89) | 56.6 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 135 | 132 | 22 | 18 | 25 | 466
  Male | 22 | 23 | 24 | 4 | 8 | 2 | 83
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 1 | 0 | 0 | 0 | 0 | 0 | 1
  ASIAN | 13 | 15 | 12 | 3 | 2 | 2 | 47
  BLACK OR AFRICAN AMERICAN | 5 | 8 | 6 | 2 | 0 | 2 | 23
  MISSING | 0 | 2 | 0 | 0 | 0 | 0 | 2
  MULTIPLE | 0 | 0 | 0 | 1 | 0 | 0 | 1
  WHITE | 137 | 133 | 138 | 20 | 24 | 23 | 475

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 20% Improvement in American College of Rheumatology Criteria (ACR20) at Week 12 Superiority Comparison With Placebo
Description: ACR20 is calculated as a 20% improvement from Baseline in Tender Joint Count 68 (TJC68) and Swollen Joint Count 66 (SJC66) and a 20% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale (VAS) with values from 0=best to 100=worst), Physician Global Assessment of Arthritis Disease Activity (PhGA) (VAS with values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS with values from 0=no pain and 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty) and an acute-phase reactant (high sensitivity C-reactive Protein mg/L (hsCRP)). For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: The analysis was performed on the ITT Set that includes all randomized participants who received at least one dose of study intervention. This population was based on the treatment the participants were randomized into. Analysis was performed using multiple imputation method to handle missing data.
Measure: Number; unit: Percentage of participants
Groups:
- Pooled Placebo: Participants between the ages of greater than or equal to (>=)18 years and less than or equal to (<=)84 years received Placebo + csDMARD administered by weekly subcutaneous injection until Week 12. The placebo arms are pooled into a single placebo arm.
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Percentage of participants | 44.8 (4.19) | 50.7 (4.12) | 57.5 (4.19) | 37.7 (5.74)
Statistical Analysis 1: Comparison: GSK3196165 90mg + csDMARD vs Pooled Placebo; The null hypothesis is that there is no difference between 90 mg dose of GSK3196165 and placebo in the proportion of participants achieving ACR20 response at Week 12 versus the alternative hypothesis that the 90 mg dose of GSK3196165 differs from placebo in the proportion of participants with ACR20 response at Week 12; Test type: Superiority; p = 0.2868, Regression, Logistic; OR and corresponding 95%CI are generated from logistic regression model adjusted for Baseline, Treatment Group, Previously Failed Medical Category; Odds Ratio (OR) = 1.38, .95% CI 2-sided [0.76 to 2.48]
Statistical Analysis 2: Comparison: GSK3196165 150mg + csDMARD vs Pooled Placebo; The null hypothesis is that there is no difference between 150 mg dose of GSK3196165 and placebo in the percentage of participants achieving ACR20 response at Week 12 versus the alternative hypothesis that the 150 mg dose of GSK3196165 differs from placebo in the percentage of participants with ACR20 response at Week 12; Test type: Superiority; p = 0.0596, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.75, .95% CI 2-sided [0.98 to 3.15]
Statistical Analysis 3: Comparison: Sarilumab 200mg + csDMARD vs Pooled Placebo; The null hypothesis is that there is no difference between 200 mg dose of Sarilumab alternating with placebo every week and placebo in the proportion of participants achieving ACR20 response at Week 12 versus the alternative hypothesis that the 200 mg dose of Sarilumab alternating with placebo every week differs from placebo in the proportion of participants with ACR20 response at Week 12; Test type: Superiority; p = 0.0049, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.34, .95% CI 2-sided [1.29 to 4.23]
Statistical Analysis 4: Comparison: GSK3196165 90mg + csDMARD vs Sarilumab 200mg + csDMARD; The null hypothesis is that there is no difference between 90 mg dose of GSK3196165 and 200 mg dose of sarilumab alternating with placebo every week in the proportion of participants achieving ACR20 response at Week 12 versus the alternative hypothesis that the 90 mg dose of GSK3196165 differs from 200 mg dose of sarilumab alternating with placebo every week in the proportion of participants with ACR20 response at Week 12; Test type: Superiority; p = 0.0293, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.59, .95% CI 2-sided [0.36 to 0.95]
Statistical Analysis 5: Comparison: GSK3196165 150mg + csDMARD vs Sarilumab 200mg + csDMARD; The null hypothesis is that there is no difference between 150 mg dose of GSK3196165 and 200 mg dose of sarilumab alternating with placebo every week in the proportion of participants achieving ACR20 response at Week 12 versus the alternative hypothesis that the 150 mg dose of GSK3196165 differs from 200 mg dose of sarilumab alternating with placebo every week in the proportion of participants with ACR20 response at Week 12; Test type: Superiority; p = 0.2308, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.75, .95% CI 2-sided [0.47 to 1.20]

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) (Versus Placebo) at Week 12
Description: Health Assessment Questionnaire-Disability Index (HAQ-DI) is a 20-question instrument that assesses the difficulty of a participant in eight domains of daily living activities: Dressing & grooming, Arising, Eating, Walking, Hygiene, Reach, Grip, Common daily activities. Overall HAQ-DI score was computed as the sum of the domain scores divided by the number of domains answered. The total possible score ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty. Higher overall score indicates greater disability. A negative change from baseline indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Scores on a scale | -0.33 (0.044) | -0.41 (0.043) | -0.46 (0.044) | -0.23 (0.061)

3. Secondary Outcome: Percentage of Participants With Clinical Disease Activity Index (CDAI) Total Score <=10 (CDAI Low Disease Activity [LDA]) at Week 12
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (TJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. Low disease activity (LDA) is achieved when CDAI total score <=10. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Percentage of participants | 20.7 (3.42) | 18.2 (3.2) | 28.1 (3.77) | 14.2 (4.15)

4. Secondary Outcome: Percentage of Participants With CDAI Total Score <=10 (CDAI LDA) at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (TJC28),Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. LDA is achieved when CDAI total score <=10.
Time Frame: Week 24
Population: The analysis was performed on all randomized participants who received study intervention from Day 01 to Week 24. Analysis was performed using multiple imputation method to handle missing data.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Percentage of participants | 31.2 | 30.1 | 42.6

5. Secondary Outcome: Percentage of Participants With CDAI Total Score <=10 (CDAI LDA) at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 4
Time Frame: Week 24
Population: The analysis was performed on all randomized participants who switched from placebo to study intervention at Week 12. Analysis was performed using multiple imputation method to handle missing data
Measure: Number; unit: Percentage of participants
Groups:
- Placebo + csDMARD and GSK3196165 90mg + csDMARD: Participants between the ages of greater than or equal to (>=)18 years and less than or equal to (<=)84 years received Placebo +csDMARD until Week 12 later switched to GSK3196165 90 mg +csDMARD administered by weekly subcutaneous injection.
- Placebo + csDMARD and GSK3196165 150mg + csDMARD: Participants between the ages of greater than or equal to (>=)18 years and less than or equal to(<=)84 years received Placebo +csDMARD until Week 12 later switched toGSK3196165 150 mg +csDMARD administered by weekly subcutaneous injection.
- Placebo + csDMARD and Sarilumab 200mg + csDMARD: Participants between the ages of greater than or equal to (>=)18 years and less than or equal to (<=)84 years received Placebo +csDMARD until Week 12 later switched toSarilumab200mg +csDMARD administered by subcutaneous injection of sarilumab every other week plus with placebo injection in the intervening weeks to maintain the blind.
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Percentage of participants | 24.0 | 42.0 | 36.1

6. Secondary Outcome: Change From Baseline in CDAI Total Score at Week 12
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (TJC28),Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. A negative CDAI total score change from baseline indicates an improvement in disease activity. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Scores on a scale | -16.87 (1.03) | -17.23 (1.018) | -20.22 (1.027) | -14.86 (1.438)

7. Secondary Outcome: Change From Baseline in CDAI Total Score at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (TJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). CDAI total score ranges from 0 to 76 with higher values representing higher disease activity.
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Scores on a scale | -20.93 (1.04) | -20.75 (1.022) | -23.22 (1.048)

8. Secondary Outcome: Change From Baseline in CDAI Total Score at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 7
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Scores on a scale | -16.84 (2.476) | -22.91 (2.439) | -20.38 (2.380)

9. Secondary Outcome: Change From Baseline in Arthritis Pain Visual Analogue Scale (VAS) at Week 12
Description: For the Arthritis Pain VAS, participants assess the severity of their current arthritis pain using a continuous visual analogue scale (VAS) with anchors at "0" (no pain) and "100" (most severe pain). A negative change from baseline indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Score on scale | -19.35 (2.127) | -21.17 (2.088) | -25.93 (2.12) | -16.73 (2.939)

10. Secondary Outcome: Change From Baseline in Arthritis Pain VAS at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: For the Arthritis Pain VAS, participants assess the severity of their current arthritis pain using a continuous visual analogue scale (VAS) with anchors at "0" (no pain) and "100" (most severe pain). A negative change from baseline indicates an improvement.
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Scores on a scale | -25.06 (2.153) | -24.31 (2.115) | -30.62 (2.141)

11. Secondary Outcome: Change From Baseline in Arthritis Pain VAS at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 10
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Scores on a scale | -16.98 (5.169) | -32.74 (5.029) | -18.60 (4.964)

12. Secondary Outcome: Percentage of Participants With CDAI Total Score <=2.8 (CDAI Remission) at Week 12
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (TJC28),Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Percentage of participants | 2.2 (1.25) | 4.3 (1.7) | 8.7 (2.38) | 0.6 (1.3)

13. Secondary Outcome: Percentage of Participants With CDAI Total Score <=2.8 (CDAI Remission) at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: as for outcome 7
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Percentage of participants | 7.9 (2.33) | 8.4 (2.32) | 8.3 (2.39)

14. Secondary Outcome: Percentage of Participants With CDAI Total Score <=2.8 (CDAI Remission) at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 7
Time Frame: Week 24
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Percentage of participants | 5.1 | 13.2 | 8.4

15. Secondary Outcome: Percentage of Participants With ACR20 at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: ACR20 is calculated as a 20% improvement from Baseline in TJC68 and SJC66 and a 20% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA), Physician Global Assessment of Arthritis Disease Activity (PhGA) (VAS values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS values from 0=no pain to 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (0=least difficulty to 3=extreme difficulty) and an acute-phase reactant (high sensitivity C-reactive Protein mg/L (hsCRP).
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Percentage of participants | 58.1 (4.18) | 60.5 (4.06) | 65.1 (4.09)

16. Secondary Outcome: Percentage of Participants With ACR20 at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 15
Time Frame: Week 24
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Percentage of participants | 61.2 | 70.7 | 55.8

17. Secondary Outcome: Percentage of Participants With 50% Improvement in American College of Rheumatology Criteria (ACR50) at Week 12
Description: ACR50 is calculated as a 50% improvement from Baseline in Tender Joint Count 68 (TJC68) and Swollen Joint Count 66 (SJC66) and a 50% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale (VAS) with values from 0=best to 100=worst), Physician Global Assessment of Arthritis Disease Activity (PhGA) (VAS with values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS with values from 0=no pain and 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty) and an acute-phase reactant (high sensitivity C-reactive Protein mg/L (hsCRP)). For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Percentage of participants | 18.2 (3.28) | 22.5 (3.47) | 25.9 (3.74) | 11.5 (3.79)

18. Secondary Outcome: Percentage of Participants With ACR50 at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: ACR50 is calculated as a 50% improvement from Baseline in TJC68 and SJC66 and a 50% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA), Physician Global Assessment of Arthritis Disease Activity (PhGA) (VAS values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS values from 0=no pain to 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (0=least difficulty to 3=extreme difficulty) and an acute-phase reactant (high sensitivity C-reactive Protein mg/L (hsCRP).
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Percentage of participants | 23.6 (3.6) | 30.1 (3.81) | 42.9 (4.25)

19. Secondary Outcome: Percentage of Participants With ACR50 at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 18
Time Frame: Week 24
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Percentage of participants | 13.1 | 41.8 | 24.0

20. Secondary Outcome: Percentage of Participants With 70% Improvement in American College of Rheumatology Criteria (ACR70) at Week 12
Description: ACR70 is calculated as a 70% improvement from Baseline in Tender Joint Count 68 (TJC68) and Swollen Joint Count 66 (SJC66) and a 70% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale (VAS) with values from 0=best to 100=worst), Physician Global Assessment of Arthritis Disease Activity (PhGA) (VAS with values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS with values from 0=no pain and 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty) and an acute-phase reactant (high sensitivity C-reactive Protein mg/L (hsCRP)). For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Percentage of participants | 5.9 (2.01) | 10.8 (2.61) | 13.3 (2.92) | 6.1 (2.93)

21. Secondary Outcome: Percentage of Participants With ACR70 at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: ACR70 is calculated as a 70% improvement from Baseline in TJC68 and SJC66 and a 70% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA), Physician Global Assessment of Arthritis Disease Activity (PhGA) (VAS values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS values from 0=no pain to 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (0=least difficulty to 3=extreme difficulty) and an acute-phase reactant (high sensitivity C-reactive Protein mg/L (hsCRP).
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Percentage of participants | 12.3 (2.81) | 13.2 (2.83) | 22.7 (3.63)

22. Secondary Outcome: Percentage of Participants With ACR70 at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 21
Time Frame: Week 24
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Percentage of participants | 4.9 | 21.4 | 12.1

23. Secondary Outcome: Percentage of Participants With Disease Activity Score Using 28 Joint Count and C-Reactive Protein (DAS28-CRP) <=3.2 (DAS28-CRP LDA) at Week 12
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-CRP scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Low disease activity (LDA) is achieved when DAS28-CRP<=3.2. A negative change from baseline in DAS28-CRP indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Percentage of participants | 17 (3.19) | 17 (3.14) | 40.1 (4.16) | 13.2 (4.06)

24. Secondary Outcome: Percentage of Participants With DAS28-CRP <=3.2 (DAS28-CRP LDA) at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-CRP scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Low disease activity (LDA) is achieved when DAS28-CRP<=3.2 . A negative change from baseline in DAS28-CRP indicates an improvement.
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Percentage of participants | 26.8 (3.75) | 24.8 (3.6) | 46.9 (4.28)

25. Secondary Outcome: Percentage of Participants With DAS28-CRP <=3.2 (DAS28-CRP LDA) at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 24
Time Frame: Week 24
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Percentage of participants | 12.5 | 43.1 | 55.9

26. Secondary Outcome: Percentage of Participants With DAS28 Erythrocyte Sedimentation Rate (ESR) <=3.2 (DAS28-ESR LDA) at Week 12
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in mm/hr), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicate less disease activity. Low disease activity (LDA) is achieved when DAS28-ESR<=3.2. A negative change from baseline in DAS28-ESR indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Percentage of participants | 13.3 (2.91) | 8.5 (2.36) | 36.2 (4.12) | 1.9 (1.86)

27. Secondary Outcome: Percentage of Participants With DAS28-ESR <=3.2 (DAS28-ESR LDA) at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in mm/hr), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicate less disease activity. Low disease activity (LDA) is achieved when DAS28-ESR<=3.2. A negative change from baseline in DAS28-ESR indicates an improvement.
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Percentage of participants | 17.4 (3.33) | 17.2 (3.23) | 45.8 (4.4)

28. Secondary Outcome: Percentage of Participants With DAS28-ESR <=3.2 (DAS28-ESR LDA) at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 27
Time Frame: Week 24
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Percentage of participants | 5.7 | 33.4 | 40.0

29. Secondary Outcome: Percentage of Participants With DAS28-CRP <2.6 (DAS28-CRP Remission) at Week 12
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-CRP scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Remission is achieved when DAS28-CRP <2.6. A negative change from baseline in DAS28-CRP indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Percentage of participants | 10.2 (2.58) | 7.2 (2.19) | 22.2 (3.51) | 1.8 (1.75)

30. Secondary Outcome: Percentage of Participants With DAS28-CRP <2.6 (DAS28-CRP Remission) at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: The DAS28-CRP arthritis is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-CRP scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Remission is achieved when DAS28-CRP <2.6. A negative change from baseline in DAS28-CRP indicates an improvement.
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Percentage of participants | 16.2 (3.14) | 13.9 (2.88) | 32.6 (4.03)

31. Secondary Outcome: Percentage of Participants With DAS28-CRP <2.6 (DAS28-CRP Remission) at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 30
Time Frame: Week 24
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Percentage of participants | 6.8 | 26.6 | 32.0

32. Secondary Outcome: Percentage of Participants With DAS28-ESR <2.6 (DAS28-ESR Remission) at Week 12
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in mm/hr), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Remission is achieved when DAS28-ESR <2.6. A negative change from baseline in DAS28-ESR indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Percentage of participants | 3.1 (1.51) | 5.7 (1.97) | 23 (3.64) | 0.7 (1.47)

33. Secondary Outcome: Percentage of Participants With DAS28-ESR <2.6 (DAS28-ESR Remission) Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in mm/hr), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Remission is achieved when DAS28-ESR <2.6. A negative change from baseline in DAS28-ESR indicates an improvement.
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Percentage of participants | 10.8 (2.74) | 8.9 (2.44) | 29.8 (4.07)

34. Secondary Outcome: Percentage of Participants With DAS28-ESR <2.6 (DAS28-ESR Remission) Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 33
Time Frame: Week 24
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Percentage of participants | 1.1 | 10.0 | 24.2

35. Secondary Outcome: Percentage of Participants With a Good/Moderate European League Against Rheumatism (EULAR) Response at Week 12
Description: DAS28-CRP and DAS28-ESR scores categorized using EULAR response criteria. Response based on the combination of current DAS28 score and the improvement in the current DAS28 score relative to baseline (Good response = DAS28 change >1.2 with current DAS28 ≤3.2; Moderate response = DAS28 change >0.6 with current DAS28 >3.2-5.1; Non-response = DAS28 change ≤0.6 and current DAS28 >5.1). For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Percentage of participants | 66.3 (4.05) | 68.4 (3.88) | 84.1 (3.14) | 62.9 (5.82)

36. Secondary Outcome: Percentage of Participants With a Good/Moderate EULAR Response at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: DAS28-CRP and DAS28-ESR scores categorised using EULAR response criteria. Response based on the combination of current DAS28 score and the improvement in the current DAS28 score relative to baseline (Good response = DAS28 change >1.2 with current DAS28 ≤3.2; Moderate response = DAS28 change >0.6 with current DAS28 >3.2-5.1; Non-response = DAS28 change ≤0.6 and current DAS28 >5.1).
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Percentage of participants | 76.3 (3.63) | 71.3 (3.77) | 86.6 (3)

37. Secondary Outcome: Percentage of Participants With a Good/Moderate EULAR Response at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 36
Time Frame: Week 24
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Percentage of participants | 73.3 | 76.7 | 83.7

38. Secondary Outcome: Percentage of Participants With ACR/EULAR Remission at Week 12
Description: Boolean-based ACR/EULAR remission is achieved if all of the following requirements are met at the same timepoint: Tender Joint Count 68 (TJC68) ≤ 1, Swollen Joint Count 66 (SJC66) ≤ 1, high sensitivity C-reactive Protein (hsCRP) ≤ 1mg/dl and patient's global assessment of disease activity (PtGA) ≤ 10. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Percentage of participants | 2 | 4 | 9 | 0

39. Secondary Outcome: Percentage of Participants With ACR/EULAR Remission at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: Boolean-based ACR/EULAR remission is achieved if all of the following requirements are met at the same timepoint: Tender Joint Count 68 (TJC68) ≤ 1, Swollen Joint Count 66 (SJC66) ≤ 1, high sensitivity C-reactive Protein (CRP) ≤ 1mg/dl and patient's global assessment of disease activity (PtGA) ≤ 10.
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Percentage of participants | 6 | 4 | 5

40. Secondary Outcome: Percentage of Participants With ACR/EULAR Remission at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 39
Time Frame: Week 24
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Percentage of participants | 1 | 1 | 1

41. Secondary Outcome: Change From Baseline in DAS28-CRP and DAS28-ESR at Week 12
Description: DAS28-CRP and DAS28-ESR are measure of RA disease activity calculated using Swollen Joint Count 28 (TJC28), Tender Joint Count 28 (TJC28), high sensitivity C-reactive Protein (hsCRP in mg/L)/Erythrocyte sedimentation rate (ESR in mm/hr (mm/hour) and patient's global assessment of disease activity (PtGA) transformed to a 0-10 scale. Total score approximate range 0-9.4, with higher scores indicating more disease activity. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Scores on a scale
  DAS28-CRP | -1.34 (0.1) | -1.42 (0.098) | -2.15 (0.1) | -1.08 (0.139)
  DAS28-ESR | -1.41 (0.109) | -1.46 (0.106) | -2.57 (0.108) | -1.06 (0.152)

42. Secondary Outcome: Change From Baseline in DAS28-CRP and DAS28-ESR at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: DAS28-CRP and DAS28-ESR are measure of RA disease activity calculated using Swollen Joint Count 28 (TJC28), Tender Joint Count 28 (TJC28), high sensitivity C-reactive Protein (hsCRP in mg/L)/Erythrocyte sedimentation rate (ESR in mm/hr (mm/hour) and patient's global assessment of disease activity (PtGA) transformed to a 0-10 scale. Total score approximate range 0-9.4, with higher scores indicating more disease activity.
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Scores on a scale
  DAS28-CRP | -1.67 (0.108) | -1.67 (0.106) | -2.38 (0.109)
  DAS28-ESR | -1.7 (0.121) | -1.68 (0.117) | -2.85 (0.121)

43. Secondary Outcome: Change From Baseline in DAS28-CRP and DAS28-ESR at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 42
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Scores on a scale
  DAS28-CRP | -1.25 (0.264) | -2.08 (0.258) | -2.15 (0.248)
  DAS28-ESR | -1.28 (0.282) | -1.94 (0.294) | -2.47 (0.266)

44. Secondary Outcome: Change From Baseline in HAQ-DI at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: Health Assessment Questionnaire-Disability Index (HAQ-DI) is a 20-question instrument that assesses the difficulty of a participant in eight domains of daily activities: Dressing & grooming, Arising, Eating, Walking, Hygiene, Reach, Grip, Common daily activities. HAQ-DI score was computed as sum of the domain scores divided by the number of domains answered. The total possible score ranges from 0=least difficulty to 3=extreme difficulty. Higher overall score indicates greater disability. A negative change from baseline indicates an improvement.
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Scores on a scale | -0.39 (0.05) | -0.45 (0.049) | -0.48 (0.05)

45. Secondary Outcome: Change From Baseline in HAQ-DI at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 44
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Scores on a scale | -0.27 (0.121) | -0.62 (0.119) | -0.32 (0.116)

46. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue at Week 12
Description: The Functional Assessment of Chronic Illness Therapy (FACIT)-fatigue is a validated patient-reported measure of 13 statements regarding the feeling of fatigue. The total score ranges from 0 to 52 with higher values representing a lower fatigue and a better quality of life. A positive change from baseline in FACIT-fatigue indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Scores on a scale | 5.5 (0.735) | 6.8 (0.724) | 7.3 (0.749) | 5.45 (1.023)

47. Secondary Outcome: Change From Baseline in FACIT-Fatigue at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: The Functional Assessment of Chronic Illness Therapy (FACIT)-fatigue is a validated patient-reported measure of 13 statements regarding the feeling of fatigue. The total score ranges from 0 to 52 with higher values representing a lower fatigue and a better quality of life. A positive change from baseline in FACIT-fatigue indicates an improvement.
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Scores on a scale | 6.55 (0.795) | 7.21 (0.777) | 7.99 (0.806)

48. Secondary Outcome: Change From Baseline in FACIT-Fatigue at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 47
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Scores on a scale | 5.48 (1.927) | 8.56 (1.852) | 7.21 (1.824)

49. Secondary Outcome: Change From Baseline in Subject-completed Medical Outcomes Study Short-Form 36 (SF-36) Physical Component Scores (PCS) at Week 12
Description: The Short-Form 36 (SF-36) is a health-related survey that assesses quality of life covering 8 domains: physical functioning, bodily pain, role limitations due to physical and emotional problems, general health, mental health, social functioning, vitality. The score for a domain was an average of the individual question scores, which were scaled 0-100; higher score represents better health. The PCS is an aggregate score derived from 4 domains (physical functioning, role-physical, bodily pain and general health) representing overall physical health. T-score scale was used for PCS with mean of 50 and SD of 10; higher score represents better health. A positive change from baseline indicates an improvement in overall physical heath. Quality Metrics software was used for scoring for SF-36. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Scores on a scale | 5.08 (0.619) | 5.03 (0.61) | 5.61 (0.627) | 3.72 (0.866)

50. Secondary Outcome: Change From Baseline in SF-36 PCS at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: The Short-Form 36 (SF-36) is a health-related survey that assesses quality of life covering 8 domains: physical functioning, bodily pain, role limitations due to physical and emotional problems, general health, mental health, social functioning, vitality. The score for a domain was an average of the individual question scores, which were scaled 0-100; higher score represents better health. The PCS is an aggregate score derived from 4 domains (physical functioning, role-physical, bodily pain and general health) representing overall physical health. T-score scale was used for PCS with mean of 50 and SD of 10; higher score represents better health. A positive change from baseline indicates an improvement in overall physical heath. Quality Metrics software was used for scoring for SF-36.
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Scores on a scale | 5.67 (0.707) | 5.5 (0.694) | 7.18 (0.71)

51. Secondary Outcome: Change From Baseline in SF-36 PCS at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 50
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Scores on a scale | 3.76 (1.687) | 8.63 (1.672) | 4.16 (1.611)

52. Secondary Outcome: Change From Baseline in SF-36 Mental Component Scores (MCS) at Week 12
Description: The Short-Form 36 (SF-36) is a health-related survey that assesses quality of life covering 8 domains: physical functioning, bodily pain, role limitations due to physical and emotional problems, general health, mental health, social functioning, vitality. The score for a domain was an average of the individual question scores, which were scaled 0-100; higher score represents better health. The MCS is an aggregated score derived from 4 domains (social functioning, vitality, mental health, and role-emotional domains) representing overall mental health. T-score scale was used for MCS with mean of 50 and SD of 10; higher score represents better health. A positive change from baseline indicates an improvement in overall mental health. Quality Metrics software was used for scoring for SF-36. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
Scores on a scale | 1.64 (0.731) | 3.45 (0.72) | 4.15 (0.744) | 1.61 (1.024)

53. Secondary Outcome: Change From Baseline in SF-36 MCS at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: The Short-Form 36 (SF-36) is a health-related survey that assesses quality of life covering 8 domains: physical functioning, bodily pain, role limitations due to physical and emotional problems, general health, mental health, social functioning, vitality. The score for a domain was an average of the individual question scores, which were scaled 0-100; higher score represents better health. The MCS is an aggregated score derived from 4 domains (social functioning, vitality, mental health, and role-emotional domains) representing overall mental health. T-score scale was used for MCS with mean of 50 and SD of 10; higher score represents better health. A positive change from baseline indicates an improvement in overall mental health. Quality Metrics software was used for scoring for SF-36.
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
Scores on a scale | 2.22 (0.772) | 3.05 (0.756) | 3.61 (0.78)

54. Secondary Outcome: Change From Baseline in SF-36 MCS at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 53
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 26 | 26 | 27
Scores on a scale | 1.44 (1.891) | 1.10 (1.855) | 2.76 (1.800)

55. Secondary Outcome: Change From Baseline in SF-36 Domain Scores at Week 12
Description: The Short-Form 36 (SF-36) is a health-related survey that assesses quality of life covering 8 domains: physical functioning, bodily pain, role limitations due to physical and emotional problems, general health, mental health, social functioning, vitality. The MCS consists of 4 domains (social functioning, vitality, mental health, and role-emotional domains) and PCS consists of 4 domains (physical functioning, role-physical, bodily pain and general health). The individual question items are first summed for each item under the various sections. Then, those domain scores are scaled between 0 to 100, where higher score represents better health. A positive change from baseline indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: The analysis was performed on the ITT Set that includes all randomized participants who received at least one dose of study intervention and for whom data available for specific parameters. This population was based on the treatment the participants were randomized into.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 143 | 148 | 138 | 71
Scores on a scale
  Bodily Pain - PCS | 17 (21.45) | 16.8 (22.2) | 19.8 (23.27) | 10.7 (21.38)
  General Health - PCS | 6.3 (15.89) | 6.7 (16.07) | 6.7 (15.69) | 4.2 (15.84)
  Role Physical - PCS | 12.94 (22.371) | 14.19 (25.155) | 13.81 (23.488) | 10.74 (19.456)
  Physical Function - PCS | 9.69 (21.423) | 14.22 (23.909) | 13.15 (24.135) | 6.55 (21.156)
  Mental Health - MCS | 4.3 (19.3) | 7.6 (16.9) | 8.2 (18.55) | 4.8 (16.31)
  Role Emotional - MCS | 5.77 (22.405) | 9.4 (25.128) | 10.93 (23.908) | 3.87 (22.219)
  Social Function - MCS | 6.99 (23.107) | 10.73 (27.51) | 11.59 (24.383) | 6.87 (27.774)
  Vitality - MCS | 9.48 (18.03) | 11.82 (19.94) | 13 (19.895) | 5.11 (18.61)

56. Secondary Outcome: Change From Baseline in SF-36 Domain Scores at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: The Short-Form 36 (SF-36) is a health-related survey that assesses quality of life covering 8 domains: physical functioning, bodily pain, role limitations due to physical and emotional problems, general health, mental health, social functioning, vitality. The MCS consists of 4 domains (social functioning, vitality, mental health, and role-emotional domains) and PCS consists of 4 domains (physical functioning, role-physical, bodily pain and general health). The individual question items are first summed for each item under the various sections. Then, those domain scores are scaled between 0 to 100, where higher score represents better health. A positive change from baseline indicates an improvement.
Time Frame: Baseline (Day 01) and Week 24
Population: The analysis was performed on all randomized participants who received study intervention from Day 01 to Week 24 and for whom data available for specific parameters.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 140 | 147 | 136
Scores on a scale
  Bodily Pain - PCS | 20.7 (22.82) | 18.5 (22.43) | 23.9 (27.29)
  General Health - PCS | 6.4 (15.25) | 6.7 (16.3) | 8.8 (17.3)
  Role Physical - PCS | 13.97 (21.332) | 15.22 (27.352) | 17.37 (26.25)
  Physical Function - PCS | 11.43 (23.714) | 16.36 (25.64) | 18.86 (24.472)
  Mental Health - MCS | 6.1 (17.16) | 8.4 (19.63) | 10 (18.71)
  Role Emotional - MCS | 5.83 (23.522) | 7.99 (28.03) | 8.88 (26.589)
  Social Function - MCS | 9.46 (25.704) | 10.37 (29.237) | 12.04 (24.599)
  Vitality - MCS | 11.29 (17.913) | 13.22 (21.245) | 16.31 (19.854)

57. Secondary Outcome: Change From Baseline in SF-36 Domain Scores at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 56
Time Frame: Baseline (Day 01) and Week 24
Population: The analysis was performed on all randomized participants who switched from placebo to study intervention at Week 12 and for whom data available for specific parameters.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 23 | 24 | 25
Scores on a scale
  Bodily Pain - PCS | 15.7 (21.91) | 20.4 (26.91) | 16.9 (23.99)
  General Health - PCS | 5.6 (14.98) | 3.4 (17.47) | 4.4 (17.20)
  Role Physical - PCS | 10.33 (21.204) | 17.19 (19.352) | 12.25 (20.530)
  Physical Function - PCS | 7.39 (19.121) | 18.75 (23.417) | 6.20 (20.630)
  Mental Health - MCS | 5.9 (14.11) | 5.2 (23.29) | 5.4 (18.54)
  Role Emotional - MCS | 7.97 (21.242) | 4.17 (28.019) | 6.67 (28.667)
  Social Function - MCS | 13.04 (23.681) | 6.25 (37.771) | 5.50 (36.279)
  Vitality - MCS | 8.42 (13.926) | 10.16 (27.263) | 11.75 (20.832)

58. Secondary Outcome: Incidence of Adverse Events (AEs), Serious Adverse Event (SAEs), Adverse Events of Special Interest (AESI)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A SAE is any untoward medical occurrence that, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity and/or can result in death.
Time Frame: Up to Week 24
Population: The analysis was performed on the Safety Set that includes all randomized participants who received at least one dose of study treatment. Pooled Placebo collected data till Week 12. Placebo + csDMARD and GSK3196165 90 mg + csDMARD, Placebo + csDMARD and GSK3196165 150 mg + csDMARD, Placebo + csDMARD and Sarilumab 200 mg or placebo + csDMARD collected data from Week 12 to 24. GSK3196165 90 mg + csDMARD, GSK3196165 150 mg + csDMARD, Sarilumab 200 mg or placebo + csDMARD collected data till Week 24
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Placebo: Participants between the ages of greater than or equal to (>=)18 years and less than or equal to (<=)84 years received Placebo + csDMARD administered by weekly subcutaneous injection until Week 12.
- Placebo + csDMARD and GSK3196165 90 mg + csDMARD: Participants received Placebo + csDMARD until Week 12 later switched to GSK3196165 90 mg + csDMARD administered by weekly subcutaneous injection.
- Placebo + csDMARD and GSK3196165 150 mg + csDMARD: Participants received Placebo + csDMARD until Week 12 later switched to GSK3196165 150 mg + csDMARD administered by weekly subcutaneous injection.
- Placebo + csDMARD and Sarilumab 200 mg + csDMARD: Participants received Placebo + csDMARD until Week 12 later switched to Sarilumab 200 mg + csDMARD administered by subcutaneous injection of sarilumab every other week plus with placebo injection in the intervening weeks to maintain the blind.
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo | Placebo + csDMARD and GSK3196165 90 mg + csDMARD | Placebo + csDMARD and GSK3196165 150 mg + csDMARD | Placebo + csDMARD and Sarilumab 200 mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156 | 79 | 24 | 25 | 26
Participants
  AE | 92 | 99 | 98 | 37 | 9 | 10 | 12
  SAE | 8 | 1 | 12 | 2 | 1 | 3 | 1
  AESI | 16 | 15 | 33 | 0 | 2 | 3 | 5

59. Secondary Outcome: Change From Baseline in Neutrophil, Lymphocyte, Platelet Count (Giga Cells Per Liter) at Week 12
Description: Blood samples was collected for the assessment of change from baseline in hematology parameters including neutrophil, lymphocyte, platelet count. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: The analysis was performed on the Safety Set that includes all randomized participants who received at least one dose of study treatment and for whom data available for specific parameters. This population was based on the treatment the participants actually received.
Measure: Mean (Standard Deviation); unit: 10^9/L (Giga cells per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 141 | 143 | 138 | 70
10^9/L (Giga cells per liter)
  Lymphocytes: number analyzed (Participants) | 141 | 143 | 137 | 70
  Lymphocytes | -0.039 (0.5089) | -0.01 (0.508) | -0.057 (0.4989) | 0.009 (0.5354)
  Neutrophils: number analyzed (Participants) | 141 | 143 | 137 | 70
  Neutrophils | -0.255 (1.5469) | -0.412 (2.0477) | -1.843 (2.1359) | -0.113 (1.4395)
  Platelets: number analyzed (Participants) | 141 | 142 | 138 | 70
  Platelets | -10.9 (56.51) | -17.3 (60.17) | -76.5 (62.76) | -10.3 (62.82)

60. Secondary Outcome: Change From Baseline in Neutrophil, Lymphocyte, Platelet Count (Giga Cells Per Liter) at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: Blood samples was collected for the assessment of change from baseline in hematology parameters including neutrophil, lymphocyte, platelet count.
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: 10^9/L (Giga cells per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 138 | 141 | 127
10^9/L (Giga cells per liter)
  Lymphocytes | -0.079 (0.5135) | 0.012 (0.5939) | -0.108 (0.52)
  Neutrophils | -0.388 (1.692) | -0.422 (1.7963) | -1.99 (2.3395)
  Platelets: number analyzed (Participants) | 135 | 141 | 127
  Platelets | -9.3 (50.96) | -9 (64.92) | -79.2 (71.13)

61. Secondary Outcome: Change From Baseline in Neutrophil, Lymphocyte, Platelet Count (Giga Cells Per Liter) at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 60
Time Frame: Baseline (Week 12) and Week 24
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: 10^9/L (Giga cells per liter)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 21 | 24 | 26
10^9/L (Giga cells per liter)
  Lymphocytes | -0.030 (0.4192) | 0.083 (0.3298) | -0.094 (0.4478)
  Neutrophils | -0.611 (1.7602) | -0.643 (1.3489) | -2.016 (2.1132)
  Platelets | -43.6 (53.10) | -12.7 (74.80) | -70.8 (82.58)

62. Secondary Outcome: Change From Baseline in White Blood Cell (WBC) Count (Giga Cells Per Liter) at Week 12
Description: Blood samples was collected for the assessment of change from baseline in hematology parameter WBC count. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: The analysis was performed on the Safety Set that includes all randomized participants who received at least one dose of study treatment. This population was based on the treatment the participants actually received.
Measure: Mean (Standard Deviation); unit: 10^9/L (Giga cells per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
10^9/L (Giga cells per liter) | -0.29 (1.753) | -0.42 (2.072) | -1.95 (2.325) | -0.09 (1.558)

63. Secondary Outcome: Change From Baseline in WBC Count (Giga Cells Per Liter) at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: Blood samples was collected for the assessment of change from baseline in hematology parameter WBC count.
Time Frame: Baseline (Day 01) and Week 24
Population: The analysis was performed on all randomized participants who received study intervention from Day 01 to Week 24.
Measure: Mean (Standard Deviation); unit: 10^9/L (Giga cells per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
10^9/L (Giga cells per liter) | -0.45 (1.851) | -0.43 (1.787) | -2.15 (2.51)

64. Secondary Outcome: Change From Baseline in WBC Count (Giga Cells Per Liter) at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: Blood samples was collected for the assessment of change from baseline in hematology parameter WBC count.
Time Frame: Baseline (Week 12) and Week 24
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: 10^9/L (Giga cells per liter)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 21 | 24 | 26
10^9/L (Giga cells per liter) | -0.66 (1.824) | -0.60 (1.452) | -2.05 (2.271)

65. Secondary Outcome: Change From Baseline in Hemoglobin Level (Grams Per Liter) Week 12
Description: Blood samples was collected for the assessment of change from baseline in hematology parameter hemoglobin level. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: g/L (Grams per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
g/L (Grams per liter) | -0.9 (8.06) | 0.3 (8.54) | 5.5 (9.19) | -2 (7.98)

66. Secondary Outcome: Change From Baseline in Hemoglobin Level (Grams Per Liter) Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: Blood samples was collected for the assessment of change from baseline in in hematology parameter hemoglobin level.
Time Frame: Baseline (Day 01) and Week 24
Population: The analysis was performed on all randomized participants who received study intervention from Day 01 to Week 24.
Measure: Mean (Standard Deviation); unit: g/L (Grams per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
g/L (Grams per liter) | -1.9 (9.05) | -1 (8.63) | 5.8 (11.07)

67. Secondary Outcome: Change From Baseline in Hemoglobin Level (Grams Per Liter) Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: Blood samples was collected for the assessment of change from baseline in in hematology parameter hemoglobin level.
Time Frame: Baseline (Week 12) and Week 24
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: g/L (Grams per liter)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 21 | 24 | 26
g/L (Grams per liter) | 3.5 (7.44) | 0.2 (10.85) | 7.0 (11.51)

68. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase (AP) Gamma-glutamyl Transferase(GGT) Levels (International Units Per Liter) at Week 12
Description: Blood samples was collected for the assessment of change from baseline in laboratory parameters including aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (AP) gamma-glutamyl transferase (GGT) levels. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: as for outcome 59
Measure: Mean (Standard Deviation); unit: IU/L (International units per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 146 | 146 | 139 | 72
IU/L (International units per liter)
  AST: number analyzed (Participants) | 144 | 145 | 137 | 70
  AST | 0.6 (10.29) | 0.7 (8.52) | 4.5 (11.43) | 0.3 (9.82)
  ALT | 0.8 (16.22) | -0.7 (12.95) | 8.1 (21.3) | -1 (10.8)
  AP: number analyzed (Participants) | 144 | 145 | 137 | 70
  AP | 0.7 (14.42) | -3 (14.94) | -15.6 (20.63) | -1 (14.57)
  GGT: number analyzed (Participants) | 144 | 145 | 137 | 70
  GGT | -0.8 (14.24) | -2.6 (15.23) | 0.6 (12.37) | -1.8 (11.46)

69. Secondary Outcome: Change From Baseline in AST, ALT, AP, GGT Levels (International Units Per Liter) at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: Blood samples was collected for the assessment of change from baseline in laboratory parameters including AST, ALT, AP, GGT levels.
Time Frame: Baseline (Day 01) and Week 24
Population: The analysis was performed on Safety Set that includes all randomized participants who received study intervention from Day 01 to Week 24 and for whom data available for specific parameters.
Measure: Mean (Standard Deviation); unit: IU/L (International units per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 141 | 145 | 129
IU/L (International units per liter)
  AST | 1.7 (7.89) | 2.1 (11.21) | 3.0 (9.29)
  ALT | 1.6 (12.73) | 1.9 (20.52) | 6.2 (12.98)
  AP | 1.8 (16.48) | -1.7 (18.76) | -14.3 (19.23)
  GGT: number analyzed (Participants) | 141 | 145 | 128
  GGT | -0.3 (13.07) | -0.3 (25.67) | 0.9 (15.73)

70. Secondary Outcome: Change From Baseline in AST, ALT, AP, GGT Levels (International Units Per Liter) at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 69
Time Frame: Baseline (Week 12) and Week 24
Population: The analysis was performed on Safety set that includes all randomized participants who switched from placebo to study intervention at Week 12 and for whom data available for specific parameters.
Measure: Mean (Standard Deviation); unit: IU/L (International units per liter)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 21 | 25 | 26
IU/L (International units per liter)
  AST: number analyzed (Participants) | 21 | 24 | 26
  AST | 2.5 (6.12) | 3.0 (9.46) | 0.9 (17.04)
  ALT | 3.3 (9.51) | 4.2 (13.08) | 3.5 (15.12)
  AP: number analyzed (Participants) | 21 | 24 | 26
  AP | 2.0 (12.25) | 1.4 (13.68) | -15.6 (18.77)
  GGT | 4.4 (13.92) | -0.8 (7.11) | -1.4 (13.04)

71. Secondary Outcome: Change From Baseline in Albumin Level (Grams Per Liter) at Week 12
Description: Blood samples was collected for the assessment of change from baseline in laboratory parameter albumin level. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: g/L (Grams per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
g/L (Grams per liter) | 0 (2.5) | 0.3 (2.38) | 1.6 (2.64) | -0.4 (2.9)

72. Secondary Outcome: Change From Baseline in Albumin Level (Grams Per Liter) at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: Blood samples was collected for the assessment of change from baseline in laboratory parameter albumin level.
Time Frame: Baseline (Day 01) and Week 24
Population: The analysis was performed on Safety set that includes all randomized participants who received study intervention from Day 01 to Week 24.
Measure: Mean (Standard Deviation); unit: g/L (Grams per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
g/L (Grams per liter) | 0.2 (2.55) | 0.2 (2.50) | 2.0 (3.16)

73. Secondary Outcome: Change From Baseline in Albumin Level (Grams Per Liter) at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: Blood samples was collected for the assessment of change from baseline in laboratory parameter albumin level.
Time Frame: Baseline (Week 12) and Week 24
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: g/L (Grams per liter)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 21 | 24 | 26
g/L (Grams per liter) | 1.6 (3.75) | 0.5 (2.43) | 1.7 (2.76)

74. Secondary Outcome: Change From Baseline in Total Bilirubin (Micromoles Per Liter) at Week 12
Description: Blood samples was collected for the assessment of change from baseline in laboratory parameter total bilirubin level. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: The analysis was performed on the ITT Set that includes all randomized participants who received at least one dose of study intervention. This population was based on the treatment the participant was randomized to.
Measure: Mean (Standard Deviation); unit: umol/L (Micromoles per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 156 | 158 | 156 | 79
umol/L (Micromoles per liter) | 0.1 (2.35) | 0.4 (3.07) | 2.3 (4.5) | 0.3 (2.64)

75. Secondary Outcome: Change From Baseline in Total Bilirubin (Micromoles Per Liter) at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: Blood samples was collected for the assessment of change from baseline in laboratory parameter bilirubin level.
Time Frame: Baseline (Day 01) and Week 24
Population: The analysis was performed on all randomized participants who received study intervention from Day 01 to Week 24.
Measure: Mean (Standard Deviation); unit: umol/L (Micromoles per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
umol/L (Micromoles per liter) | 0.1 (2.06) | 0.2 (2.70) | 2.5 (4.11)

76. Secondary Outcome: Change From Baseline in Total Bilirubin (Micromoles Per Liter) at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: Blood samples was collected for the assessment of change from baseline in laboratory parameter bilirubin level.
Time Frame: Baseline (Week 12) and Week 24
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: umol/L (Micromoles per liter)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 21 | 25 | 26
umol/L (Micromoles per liter) | 0.8 (1.97) | -0.2 (3.17) | 1.1 (3.39)

77. Secondary Outcome: Change From Baseline in Total Cholesterol (Millimoles Per Liter) at Week 12
Description: Blood samples was collected for the assessment of change from baseline in lipid profile of total cholesterol levels. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: Blood samples were collected at indicated time points as per schedule of assessment in the protocol. The Objectives and Endpoints section incorrectly states that Change from baseline in key laboratory parameters at Week 12 was a secondary objective, however for the lipid panel, there is no corresponding time point in the schedule of assessment. Consequently, the only objective that can be assessed for the lipid panel is Week 4 and not at Week 12.
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

78. Secondary Outcome: Change From Baseline in Total Cholesterol (Millimoles Per Liter) at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: Blood samples was collected for the assessment of change from baseline in lipid profile of total cholesterol levels.
Time Frame: Baseline (Day 01) and Week 24
Population: The analysis was performed on all randomized participants who received study intervention from Day 01 to Week 24.
Measure: Mean (Standard Deviation); unit: mmol/L (Millimoles per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
mmol/L (Millimoles per liter) | 0.053 (1.0158) | 0.061 (0.7881) | 0.445 (0.8863)

79. Secondary Outcome: Change From Baseline in Total Cholesterol (Millimoles Per Liter) at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: Blood samples was collected for the assessment of change from baseline in lipid profile of total cholesterol levels.
Time Frame: Baseline (Week 12) and Week 24
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: mmol/L (Millimoles per liter)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 20 | 23 | 25
mmol/L (Millimoles per liter) | 0.126 (0.8456) | -0.006 (0.7593) | 0.731 (0.8654)

80. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: Low-density Lipoprotein (LDL) Cholesterol, High-density Lipoprotein (HDL) Cholesterol (Millimoles Per Liter) at Week 12
Description: Blood samples was collected for the assessment of change from baseline in fasting lipid profile including LDL cholesterol, HDL cholesterol levels. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: as for outcome 77
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

81. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: LDL Cholesterol, HDL Cholesterol (Millimoles Per Liter) at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: Blood samples was collected for the assessment of change from baseline in fasting lipid profile including LDL cholesterol, HDL cholesterol levels.
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: mmol/L (Millimoles per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 140 | 142 | 125
mmol/L (Millimoles per liter)
  HDL Cholesterol, Direct | 0.044 (0.2523) | 0.051 (0.2931) | 0.063 (0.2784)
  LDL Cholesterol: number analyzed (Participants) | 138 | 140 | 125
  LDL Cholesterol | -0.026 (0.8577) | 0.021 (0.6769) | 0.334 (0.7472)

82. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: LDL Cholesterol, HDL Cholesterol (Millimoles Per Liter) at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 81
Time Frame: Baseline (Week 12) and Week 24
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: mmol/L (Millimoles per liter)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 20 | 23 | 25
mmol/L (Millimoles per liter)
  HDL Cholesterol, Direct | 0.049 (0.2578) | 0.000 (0.2511) | 0.107 (0.3202)
  LDL Cholesterol | 0.041 (0.7034) | 0.006 (0.6861) | 0.513 (0.6822)

83. Secondary Outcome: Change From Baseline in Fasting Lipid Profile Triglycerides (Millimoles Per Liter) at Week 12
Description: Blood samples was collected for the assessment of change from baseline in fasting lipid profile triglycerides levels. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: as for outcome 77
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

84. Secondary Outcome: Change From Baseline in Fasting Lipid Profile Triglycerides (Millimoles Per Liter) at Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: Blood samples was collected for the assessment of change from baseline in fasting lipid profile triglycerides levels.
Time Frame: Baseline (Day 01) and Week 24
Population: The analysis was performed on all randomized participants who received study intervention from Day 01 to Week 24.
Measure: Mean (Standard Deviation); unit: mmol/L (Millimoles per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156
mmol/L (Millimoles per liter) | 0.075 (0.5799) | -0.038 (0.5519) | 0.103 (0.7552)

85. Secondary Outcome: Change From Baseline in Fasting Lipid Profile Triglycerides (Millimoles Per Liter) at Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: Blood samples was collected for the assessment of change from baseline in fasting lipid profile triglycerides levels.
Time Frame: Baseline (Week 12) and Week 24
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: mmol/L (Millimoles per liter)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 20 | 23 | 25
mmol/L (Millimoles per liter) | 0.072 (0.4498) | -0.024 (0.5497) | 0.243 (0.8130)

86. Other Pre Specified Outcome: Change From Baseline 4-beta-hydroxy Cholesterol, Cholesterol at (Millimoles Per Liter) Week 12
Description: Blood samples was collected for the assessment of change from baseline in lipid profile parameter including 4-beta-hydroxycholesterol, cholesterol levels. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 01) and Week 12
Population: as for outcome 59
Measure: Mean (Standard Deviation); unit: mmol/L (Millimoles per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo
Number analyzed (Participants) | 139 | 141 | 134 | 71
mmol/L (Millimoles per liter)
  4-Beta-Hydroxycholesterol | 0.9897 (0.81483) | 1.0156 (0.57323) | 1.1148 (0.56873) | 1.0913 (1.03027)
  Cholesterol: number analyzed (Participants) | 129 | 136 | 126 | 69
  Cholesterol | 58.5438 (13.25606) | 59.1757 (14.83734) | 64.3791 (15.12089) | 58.6880 (14.62446)

87. Other Pre Specified Outcome: Change From Baseline 4-beta-hydroxy Cholesterol, Cholesterol at (Millimoles Per Liter) Week 24 for Treatment Arms That Started Study Intervention From Day 1
Description: Blood samples was collected for the assessment of change from baseline in lipid profile parameter including 4-beta-hydroxycholesterol, cholesterol levels.
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: mmol/L (Millimoles per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 136 | 139 | 123
mmol/L (Millimoles per liter)
  4-Beta-Hydroxycholesterol | 0.9766 (0.45665) | 1.0064 (0.58945) | 1.1925 (0.57339)
  Cholesterol: number analyzed (Participants) | 133 | 137 | 121
  Cholesterol | 59.1937 (14.12055) | 58.9174 (15.00108) | 65.2270 (14.70946)

88. Other Pre Specified Outcome: Change From Baseline 4-beta-hydroxy Cholesterol, Cholesterol at (Millimoles Per Liter) Week 24 for Placebo Switched Arms That Started Study Intervention From Week 12
Description: as for outcome 87
Time Frame: Baseline (Week 12) and Week 24
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: mmol/L (Millimoles per liter)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 20 | 23 | 24
mmol/L (Millimoles per liter)
  4-Beta-Hydroxycholesterol | 1.0180 (0.42435) | 0.9467 (0.29136) | 1.3897 (1.31589)
  Cholesterol: number analyzed (Participants) | 18 | 22 | 24
  Cholesterol | 56.7570 (13.92076) | 62.4284 (13.72140) | 68.7768 (17.39453)

89. Secondary Outcome: Number of Participants With National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) >=Grade 3 Hematological/Clinical Chemistry Abnormalities for Treatment Arms That Started Study Intervention From Day 1
Description: Number of participants who reported NCI-CTCAE Grade 3 or higher for hematological and clinical chemistry abnormalities were summarized.
Time Frame: Up to Week 24
Population: The analysis was performed on the randomized participants who received at least one dose of study treatment and for whom data available for specific parameters. Pooled Placebo collected data till Week 12. Placebo+csDMARD and GSK3196165 90mg+csDMARD, Placebo+csDMARD and GSK3196165 150mg+csDMARD, Placebo+csDMARD and Sarilumab 200mg or placebo+csDMARD collected data from Week 12 to 24. GSK3196165 90mg+csDMARD, GSK3196165 150mg+csDMARD, Sarilumab 200mg or placebo+csDMARD collected data till Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo | Placebo + csDMARD and GSK3196165 90mg + csDMARD | Placebo + csDMARD and GSK3196165 150mg + csDMARD | Placebo + csDMARD and Sarilumab 200mg + csDMARD
Number analyzed (Participants) | 155 | 156 | 153 | 78 | 24 | 25 | 26
Participants
  Alanine aminotransferase increased, Total, Grade 3 | 1 | 2 | 1 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased, Total, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased, Total, Grade 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased, Total, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased, Total, Grade 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Blood bilirubin increased, Total, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased, Total, Grade 3 | 6 | 1 | 2 | 0 | 0 | 0 | 0
  Lymphocyte count decreased, Total, Grade 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Lymphocyte count increased, Total, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased, Total, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil count decreased, Total, Grade 3 | 2 | 1 | 10 | 0 | 1 | 1 | 2
  Neutrophil count decreased, Total, Grade 4 | 1 | 1 | 4 | 0 | 0 | 0 | 0
  Platelet count decreased, Total, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased, Total, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0

90. Secondary Outcome: Concentrations of Granulocyte-macrophage Colony Stimulating Factor (GM-CSF) Autoantibody
Description: Blood samples were collected for markers which may influence rheumatoid arthritis. Concentrations of GM-CSF autoantibodies was determined.
Time Frame: At baseline
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: ug/L (microgram per liter)
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Placebo + csDMARD and GSK3196165 90 mg + csDMARD | Placebo + csDMARD and GSK3196165 150 mg + csDMARD | Placebo + csDMARD and Sarilumab 200 mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156 | 26 | 26 | 27
ug/L (microgram per liter) | 334.008 (823.7538) | 417.378 (1632.7755) | 250.015 (671.9296) | 237.1 (357.4074) | 330.527 (496.9961) | 142.446 (169.6796)

91. Secondary Outcome: Number of Participants With Anti-GSK3196165 Antibodies
Description: Blood samples were collected for anti-GSK3196165 antibodies detection assay using tiered testing schema: screening, confirmation and titration steps was used for immunogenicity analysis.
Time Frame: Up to Week 24
Population: as for outcome 62
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Placebo + csDMARD and GSK3196165 90 mg + csDMARD | Placebo + csDMARD and GSK3196165 150 mg + csDMARD | Placebo + csDMARD and Sarilumab 200 mg + csDMARD
Number analyzed (Participants) | 156 | 158 | 156 | 26 | 26 | 27
Participants | 4 | 2 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were collected from the start of study intervention. The Pooled Placebo collected during the timeframe Week 0 to Week 12. Placebo + csDMARD and GSK3196165 90 mg + csDMARD, Placebo + csDMARD and GSK3196165 150 mg + csDMARD, Placebo + csDMARD and Sarilumab 200 mg or placebo + csDMARD collected during the timeframe Week 12 to Week 24. GSK3196165 90 mg + csDMARD, GSK3196165 150 mg + csDMARD, Sarilumab 200 mg or placebo + csDMARD collected during the timeframe Week 0 to Week 24.
Arm/Group | GSK3196165 90mg + csDMARD | GSK3196165 150mg + csDMARD | Sarilumab 200mg + csDMARD | Pooled Placebo | Placebo + csDMARD and GSK3196165 90 mg + csDMARD | Placebo + csDMARD and GSK3196165 150 mg + csDMARD | Placebo + csDMARD and Sarilumab 200 mg + csDMARD
All-Cause Mortality (participants affected / at risk) | 1/156 | 0/158 | 1/156 | 0/79 | 0/24 | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 8/156 | 1/158 | 12/156 | 2/79 | 1/24 | 3/25 | 1/26
Other Adverse Events (participants affected / at risk) | 25/156 | 32/158 | 41/156 | 5/79 | 1/24 | 4/25 | 6/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3196165 90mg + csDMARD (N=156) | GSK3196165 150mg + csDMARD (N=158) | Sarilumab 200mg + csDMARD (N=156) | Pooled Placebo (N=79) | Placebo + csDMARD and GSK3196165 90 mg + csDMARD (N=24) | Placebo + csDMARD and GSK3196165 150 mg + csDMARD (N=25) | Placebo + csDMARD and Sarilumab 200 mg + csDMARD (N=26)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drowning (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellar hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3196165 90mg + csDMARD (N=156) | GSK3196165 150mg + csDMARD (N=158) | Sarilumab 200mg + csDMARD (N=156) | Pooled Placebo (N=79) | Placebo + csDMARD and GSK3196165 90 mg + csDMARD (N=24) | Placebo + csDMARD and GSK3196165 150 mg + csDMARD (N=25) | Placebo + csDMARD and Sarilumab 200 mg + csDMARD (N=26)
Alanine aminotransferase increased (Investigations) | 2 (2) | 6 (6) | 10 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 10 (10) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 9 (17) | 10 (11) | 17 (35) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 11 (12) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 8 (10) | 8 (9) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Latent tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT04134728/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT04134728/SAP_001.pdf